CLINICAL TRIAL: NCT02426606
Title: The Love of Lentils (LoL) Study: The Effects of Acute Consumption of Common Lentil Varieties on Post-prandial Blood Glucose and Insulin Levels in Healthy Adult
Brief Title: Effects of Lentil Consumption on Post-prandial Blood Glucose and Insulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government); Pulse Canada (Other); Saskatchewan Pulse Growers (Other)
Responsible Party: Principal Investigator, Alison Duncan, Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 14SE012
Record Dates: First submitted 2015-04-16; First posted 2015-04-27 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: Lentils; Post-prandial; Glycemic response; Insulin response; Diabetes; Mixed meal; Glycemia; Slowly digestible starch; Post-prandial glycemia
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- White bread (Experimental)
  Interventions: Other: Various lentil varieties (varying in slow digested starch content)
- Lentil 1 + white rice (Experimental)
  Interventions: Other: Various lentil varieties (varying in slow digested starch content)
- Lentil 2 + white rice (Experimental)
  Interventions: Other: Various lentil varieties (varying in slow digested starch content)
- Lentil 3 + white rice (Experimental)
  Interventions: Other: Various lentil varieties (varying in slow digested starch content)
- White rice (Experimental)
  Interventions: Other: Various lentil varieties (varying in slow digested starch content)
- Lentil 1 + potato (Experimental)
  Interventions: Other: Various lentil varieties (varying in slow digested starch content)
- Lentil 2 + potato (Experimental)
  Interventions: Other: Various lentil varieties (varying in slow digested starch content)
- Lentil 3 + potato (Experimental)
  Interventions: Other: Various lentil varieties (varying in slow digested starch content)
- Potato (Experimental)
  Interventions: Other: Various lentil varieties (varying in slow digested starch content)

INTERVENTIONS:
Other: Various lentil varieties (varying in slow digested starch content) — Randomized, cross-over block design.
  Comparison of glycemic and insulinemic responses following meals composed of:
  * white rice or white rice combined with 1 of 3 different lentil varieties or
  * white potato or white potato combined with 1 of 3 different lentil varieties
  Participants with be assigned to either the white rice or white potato group. Meals will provide 50g available carbohydrate (AC). In meals containing lentils, whole cooked lentils will provide 25g AC either white rice or white potato will provide 25g AC.
  Meals will be randomly consumed across 6 study visits, with 2 white bread control meals (one of which will take place on the first visit).

SUMMARY:
The purpose of this study is to assess the effects of consuming various lentil varieties in mixed-meals (containing either white rice or white potato) on post-prandial blood glucose and insulin as compared to white rice or white potato alone.

DETAILED DESCRIPTION:
Eligible participants will undergo a total of 6 study visits. During each visit, a fasted blood sample will be taken by fingerprick, and approximately 500µL of blood will be dripped into a collection tube. The participant will then consume a meal of either: white bread, white rice (or white potato), or white rice with lentils (or white potato with lentils). White bread will be consumed on the first study visit and the rest of the meals will take place in random order in the visits following. Each meal will provide a total of 50g available carbohydrate. Six more blood samples will be taken by fingerprick at 15, 30, 45, 60, 90 and 120 minutes after the beginning of the meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Age 18-40 years
* BMI 20-30 kg/m2

Exclusion Criteria:

* Tobacco use
* Pregnant or breastfeeding
* Fasting blood glucose ≥ 7.0 mmol/L
* Any major medical condition including a history of AIDS or hepatitis
* Medical or surgical event requiring hospitalization within 3 months of randomization
* Any medications except a stable dose (3 months) of oral contraceptives, blood pressure or statin medications
* Blood pressure >140/90 mm Hg
* Natural health products (NHPs) used for glycemic control
* Probiotic supplements
* Dietary fibre supplements
* Consumption of >4 servings of pulses per week
* Food allergy or non-food life threatening allergy
* Shift workers
* Alcohol consumption >14 drinks/week or >4 drinks/sitting
* Recent or intended significant weight loss or gain (>4 kg in previous 3 months)
* Elite athletes

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose | Acute- 2 hours following meal
  Different meals will be consumed on separate occasions over 3-6 week period.
Postprandial blood insulin | Acute- 2 hours following meal
  Different meals will be consumed on separate occasions over 3-6 week period.

CONTACTS AND LOCATIONS:
Overall Officials: Alison M Duncan, Ph.D, R.D, Principal Investigator — University of Guelph
Locations (1):
- Human Nutraceutical Research Unit, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moravek D, Duncan AM, VanderSluis LB, Turkstra SJ, Rogers EJ, Wilson JM, Hawke A, Ramdath DD. Carbohydrate Replacement of Rice or Potato with Lentils Reduces the Postprandial Glycemic Response in Healthy Adults in an Acute, Randomized, Crossover Trial. J Nutr. 2018 Apr 1;148(4):535-541. doi: 10.1093/jn/nxy018. PMID 29659967